CLINICAL TRIAL: NCT05598866
Title: Correlation Between the Serum Chloride Levels and the Anion Gap Values in the Initial Fluid Resuscitation in DKA Patients and Its Relation to Outcome
Brief Title: Correlation Between Serum Chloride and Anion Gap Levels in DKA Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mervat Mokhles Fathi Sayed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mervat Mokhles Fathi Sayed, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Serum chloride in DKA
Record Dates: First submitted 2022-08-19; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Correlation Between Serum Chloride and Anion Gap in DKA Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
2.2 Aim(s) of the Research (50 words max):

1. To examine the description and correlation of changes in the serum chloride levels and changes in the anion gap values before and after fluid resuscitation in patients with DKA and to examine the description and correlation of changes in the serum chloride.
2. relation of serum chloride and outcome in patients with DKA

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is one of the most serious and acute complications of diabetes. DKA is a significant contributor to mortality, costs, and poor quality of life.

The total incidence of DKA tends to increase, mainly due to an increase in type 2 diabetes cases and obesity.

DKA consists of the biochemical triad of hyperglycemia, ketonemia, and metabolic acidosis resulting from absolute or relative insulin deficiency and an increase in counter-regulatory hormones. These life-threatening consequences produce severe body water deficit, the accumulation of ketone bodies, and electrolyte disturbances.

Hyperglycemia develops because of three processes: increased gluconeogenesis, accelerated glycogenolysis, and impaired glucose utilization by peripheral tissues. The hyperglycemia will lead to glycosuria and osmotic diuresis, resulting in hyperosmolar intracellular dehydration.

In DKA, fluid deficits may be up to 10% of total body weight and electrolyte deficits in the body, one of which is chloride.

In DKA, lipolysis resulting in high circulating levels of free fatty acids may occur. These free fatty acids are taken up by the liver and oxidized to ketone bodies. Excessive production of ketone bodies in the anionic form can cause high plasma anion gap. Ketone bodies are relatively strong acids that dissociate at physiologic pH. The dissociation in the form of H+ ions will be buffered by bicarbonate. When the plasma bicarbonate concentrations decrease, a high anion gap acidosis metabolic (HAGMA) develops. The anion gap calculation formula is [Na+ (Cl-+ HCO3)]. Based on diagnostic criteria, the anion gap value in DKA >10. The increased anion gap is a predictor of metabolic acidosis, and the degree of metabolic acidosis can be estimated by the size of the anion gap. Initial management of adult patients with DKA is rehydration with normal saline fluid (0.9% NaCl) intravenously and insulin administration (when the serum potassium levels <3.3 mEq/L). The initial dose of normal saline infusion is 15-20 mL/kg/hour over the first hour.

Subsequent amount of fluid given depends on the hydration status, hemodynamic conditions, and electrolyte levels. Electrolyte levels are monitored after 2 hours of initial fluid resuscitation.

The goals of rapid rehydration are to improve the circulatory volume and tissue perfusion, clear ketone bodies, and correct electrolyte imbalances. Normal saline contains 154 mEq/L chloride and 154 mEq/L sodium.

The chloride concentration of saline is higher than that of human plasma (97-107 mEq/L).

Normal saline (0.9% sodium chloride) is a low-cost and easy-to-find crystalloid fluid which becomes fluid choice by doctors in some cases. However, normal saline is now under observation due to concerns about hyperchloremic metabolic acidosis, oliguria, prolonged acidosis, and coagulopathy. Consistent data are found regarding increased serum chloride levels associated with complications of acidosis, AKI, or electrolyte disturbances after being given at least 2 liters of normal saline. An increase in the chloride levels is not counterbalanced by an increase in the bicarbonate ion concentrations in plasma. Although the anion gap values decrease, acidosis still occurs. Thus, normal anion gap metabolic acidosis (NAGMA) or hyperchloremic acidosis arises.

Blood glucose level <200 mg/dL, serum bicarbonate level >15 mEq/L, pH >7.3, and normal anion gap are recovery signs of DKA.12 causes of hyperchloremia include: Gastrointestinal problems, such as vomiting or diarrhea. heat exposure, Diabetes insipidus, Some medications, particularly hormones as estrogens, diuretics, corticosteroids,and certain,chemotherapy Starvation due to eating disorders, severe malnourishment, or problems absorbing nutrients from food.

Addison's disease, diabetes insipidus,burns, kidney disease, kidney failure, and renal tubular acidosis

Hypochloremia can be caused by:

Diarrhea Vomiting Excessive sweating Kidney problems Chronic respiratory acidosis, Syndrome of inappropriate antidiuretic hormone excretion (SIADH), Metabolic alkalosis, Use of certain medications like corticosteroids, diuretics, laxatives, and bicarbonates

ELIGIBILITY:
Inclusion Criteria:

* any patients admitted to intensive care unit, critical care unit in Assuit university from 15 yrs to 70
* Blood glucose level >250 mg/dl ( normal 70-100)
* Ph<7.3 ( normal PH 7.35- 7.45)Hco3<15 m mol/litre ( normal HCO3 22-26)
* Serum chloride before resucitation <107m mol/litre (normal 96- 106)
* Urea <6.5 m mol/litre
* S.create <120 m mol/litre

Exclusion Criteria:

* Patients receiving chemotherapy, diuretics, corticosteroids, laxatives
* Patients diagnosed to have Addison disease
* Patients with chronic kidney disease and acute kidney injury, end stage renal disease, renal tubular acidosis
* Patients with malabsorpion syndrome ( celiac disease, crohn's , celiac disease )
* Patients with chronic respiratory acidosis (asthma, COPD, pulmonary fibrosis, neuromuscular disorders)
* Patients with diarrhea

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: any patients admitted to intensive care unit, critical care unit in Assuit university from……to……..
  * Blood glucose level >250 mg/dl ( normal 70-100)
  * Ph<7.3 ( normal PH 7.35- 7.45)
  * Hco3<15 m mol/litre ( normal HCO3 22-26)
  * Serum chloride before resucitation <107m mol/litre (normal 96- 106)
  * Urea <6.5 m mol/litre
  * S.create <120 m mol/litre
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
1-Change in serum chloride levels before and after fluid resucitation in DKA patients. 2- change in anion gap level before and after fluid resuscitation in DKA patients. | 2 years
  1. change in serum chloride level before and after fluid resuscitation in DKA patients.
  2. change in anion gap level before and after fluid resuscitation in DKA patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided